CLINICAL TRIAL: NCT00992823
Title: Iron Supplementation to Reduce Preschoolers Anemia: Comparison Between Intermittent and Cyclic Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Jose do Rio Preto Medical School (Other)
Responsible Party: Geraldo Gaspar Paes Leme Coutinho, Sao Jose do Rio Preto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0708/2006
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Anemia
Keywords: Iron; anemia; supplementation; preschoolers; prevalence; preschoolers children from public day care centers
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1:iron weekly supplementation (Active Comparator)
  Interventions: Drug: iron supplementation
- Group 2: cycle supplementation (Active Comparator): two 5-month cycles, each cycle consisting of one month of supplementation (20 workdays) and four months without supplementation.
  Interventions: Biological: iron supplementation

INTERVENTIONS:
Drug: iron supplementation — 40 doses of 30 mg of ferrous sulfate during a 10-month intervention period
  Arms: Group 1:iron weekly supplementation
Biological: iron supplementation — supplementation in two 5-month cycles, each cycle consisting of one month of supplementation (20 workdays) and four months without supplementation.
  Arms: Group 2: cycle supplementation

SUMMARY:
Aim: To evaluate the efficacy of iron supplements given at intervals corresponding to the mean life of red blood cells compared to weekly supplementation, in reducing the prevalence of preschool anemia.

Method: Ninety-nine children from public day care centers with ages from 24 to 59 months old were randomly divided into two groups. All the children received 40 doses of 30 mg of ferrous sulfate during a 10-month intervention period. Group 1 received once weekly supplementation and Group 2 received supplementation in two 5-month cycles, each cycle consisting of one month of supplementation (20 workdays) and four months without supplementation.

DETAILED DESCRIPTION:
The prevalence of anemia after the supplementation regimens reduced from 20.20% to 5.05% (P < 0.0005); the reduction was not significantly different between the two groups (P = 0.35). The mean hemoglobin concentration increased in both groups (Group 1: 0.27 g/dL; P < 0.016 and Group 2: 0.47 g/dL; P < 0.0005) without significant differences between the groups (P = 0.17).

ELIGIBILITY:
Inclusion Criteria:

* The participants of the study were children with ages ranging from 24 to 59 months old that attended four local public day care centers

Exclusion Criteria:

* Presence of infection or reported infections within two weeks prior to the intervention
* Anemia lower than 7.0 g/dL and children taking medications containing ferrous sulfate

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2006-03; Primary Completion 2007-02 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Initial and final blood hemoglobin concentration | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M Cury, MDPhD, Study Director — FAMEP; Geraldo PL Coutinho, MD, Principal Investigator — Sao Jose do Rio Preto Medical School
Locations (1):
- Public Day Care Centers, Badi Bassit, São Paulo, Brazil

REFERENCES:
- [Derived] Coutinho GG, Cury PM, Cordeiro JA. Cyclical iron supplementation to reduce anemia among Brazilian preschoolers: a randomized controlled trial. BMC Public Health. 2013 Jan 10;13:21. doi: 10.1186/1471-2458-13-21. PMID 23305566